CLINICAL TRIAL: NCT05602818
Title: A Phase 1, Randomized, Double-Blind, Double-Dummy, Active- and Placebo-Controlled, 5-Way Crossover Study Evaluating the Abuse Potential of Soticlestat (TAK-935) in Healthy Adult Nondependent Recreational Drug Users With Central Nervous System Depressant Experience
Brief Title: A Study of Soticlestat in Healthy Adult Nondependent Recreational Drug Users With Central Nervous System (CNS) Depressant Experience
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: TAK-935-1012
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — soticlestat; Alprazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Soticlestat 300 mg (Experimental): Participants will receive a single oral dose of soticlestat 300 milligrams (mg).
  Interventions: Drug: Soticlestat 300 mg
- Soticlestat 600 mg (Experimental): Participants will receive a single oral dose of soticlestat 600 mg.
  Interventions: Drug: Soticlestat 600 mg
- Soticlestat 900 mg (Experimental): Participants will receive a single oral dose of soticlestat 900 mg.
  Interventions: Drug: Soticlestat 900 mg
- Alprazolam 2 mg (Active Comparator): Participants will receive a single oral dose of over encapsulated alprazolam 2 mg.
  Interventions: Drug: Alprazolam
- Placebo (Placebo Comparator): Participants will receive a single oral dose of matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Soticlestat 300 mg — Administered orally.
  Arms: Soticlestat 300 mg
Drug: Soticlestat 600 mg — Administered orally.
  Arms: Soticlestat 600 mg
Drug: Soticlestat 900 mg — Administered orally.
  Arms: Soticlestat 900 mg
Drug: Alprazolam — Administered orally.
  Arms: Alprazolam 2 mg
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main aim is to evaluate the relative abuse potential of soticlestat in healthy adults who has used central nervous system (CNS) depressants for recreational nontherapeutic reasons.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat. Soticlestat is being tested in healthy participants. This study will assess the relative abuse potential of soticlestat compared to alprazolam and placebo in healthy adult, nondependent recreational drug users with CNS depressant experience. The study will enroll approximately 110 participants. Participants will be randomly (by chance, like flipping a coin) assigned to treatments of the study.

Treatment order will remain undisclosed to the participants and study doctor (unless there is an urgent medical need). This single center trial will be conducted in the United States. Participants will be followed up for up to 7 days after the last dose of study drug for a follow-up assessment. The overall time to participate in this study is approximately 11 weeks.

ELIGIBILITY:
Inclusion Criteria

1. Healthy as determined by the investigator.
2. Current CNS depressant user who has used CNS depressants (example, benzodiazepines, barbiturates, zolpidem, eszopiclone, zopiclone, propofol/fospropofol, gamma-hydroxybutyrate) for recreational, nontherapeutic reasons at least 10 times in their lifetime and at least once in the 12 weeks prior to screening. Participant must also have recreational experience with at least 1 other drug class associated with abuse (example, opioids, stimulants, cannabinoids, hallucinogens, dissociatives) at least 10 times in their lifetime.
3. Body mass index (BMI) of 18.5 to 35.0 kilogram per square meter (kg/m^2), inclusive, and a minimum body weight of 50.0 Kilogram (kg) at screening.

Exclusion Criteria

1. Self-reported history of drug or alcohol dependence (within the past 1 year, except caffeine or nicotine, prior to the screening visit).
2. Positive alcohol breathalyzer or urine drug screen (UDS) for substances of abuse at admission, excluding tetrahydrocannabinol (THC).
3. Heavy smoker or user of other types of nicotine products (greater than [>] 20 cigarettes equivalent per day).
4. Unable to abstain from smoking for at least 2 hours before and at least 8 hours after dosing.
5. Consumes excessive amounts, defined as greater than 4 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Altasciences, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://classic.clinicaltrials.gov/ct2/bye/kQoPWwoRrXS90dhzuQ7gkdoPSQ7GvwSxWB7mz6hjuBc9mX-gWi7PxX7PzihGedY9kRh8EB76k6NjLK7jWKCtOscz5PNzvihHSsD8LVp8SRzP3DSWxRF8mRCtaRp8SRp8LPt/3HhqJdcyWB7zunhLZwN8JQ7xNd-ymB1PedcOJdcOJihkznogWi7PxXY30dhz0QS3l61yzXc9unoPlQ1RJdhzuQSO

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 15 November 2022 to 07 July 2023. A total of 100 participants participated in the Qualification Phase, of which 69 met the qualification criteria, out of which 68 enrolled in the treatment phase and were randomized to 1 of the 10 sequences of the Treatment Phase.
Pre-assignment Details: Participants entered a Qualification Phase to determine if they were able to discriminate the drug effects of the positive control, alprazolam, when compared with placebo. Only participants who could discriminate the drug effects of the positive control were randomized into one of the 10 sequences of Treatment Phase (ABECD, BCADE, CDBEA, DECAB, EADBC, DCEBA, EDACB, AEBDC, BACED or CBDAE) to receive soticlestat, alprazolam or placebo.
Groups:
- Qualification Phase: Sequence 1: All participants received:
  Day 1: Alprazolam 2 milligrams (mg), Day 2: Alprazolam matching placebo. Orally with a 4-day washout between Qualification Phase and Treatment Phase.
- Qualification Phase: Sequence 2: All participants received:
  Day 1: Alprazolam matching placebo, Day 2: Alprazolam 2 mg. Orally with a 4-day washout between Qualification Phase and Treatment Phase.
- Treatment Phase, Sequence 1: ABECD: All participants received:
  Period 1: Soticlestat 300 milligrams (mg) (Treatment A), Period 2: Soticlestat 600 mg (Treatment B), Period 3: Placebo (Treatment E), Period 4: Soticlestat 900 mg (Treatment C), Period 5: Alprazolam 2 mg (Treatment D). Orally with a 7-day washout between doses.
- Treatment Phase, Sequence 2: BCADE: All participants received:
  Period 1: Soticlestat 600 mg (Treatment B), Period 2: Soticlestat 900 mg (Treatment C), Period 3: Soticlestat 300 mg (Treatment A), Period 4: Alprazolam 2 mg (Treatment D), Period 5: Placebo (Treatment E). Orally with a 7-day washout between doses.
- Treatment Phase, Sequence 3: CDBEA: All participants received:
  Period 1: Soticlestat 900 mg (Treatment C), Period 2: Alprazolam 2 mg (Treatment D), Period 3: Soticlestat 600 mg (Treatment B), Period 4: Placebo (Treatment E), Period 5: Soticlestat 300 mg (Treatment A). Orally with a 7-day washout between doses.
- Treatment Phase, Sequence 4: DECAB: Period 1: Alprazolam 2 mg (Treatment D), Period 2: Placebo (Treatment E), Period 3: Soticlestat 900 mg (Treatment C), Period 4: Soticlestat 300 mg (Treatment A), Period 5: Soticlestat 600 mg (Treatment B). Orally with a 7-day washout between doses.
- Treatment Phase, Sequence 5: EADBC: All participants received:
  Period 1: Placebo (Treatment E), Period 2: Soticlestat 300 mg (Treatment A), Period 3: Alprazolam 2 mg (Treatment D), Period 4: Soticlestat 600 mg (Treatment B), Period 5: Soticlestat 900 mg (Treatment C). Orally with a 7-day washout between doses.
- Treatment Phase, Sequence 6: DCEBA: All participants received:
  Period 1: Alprazolam 2 mg (Treatment D), Period 2: Soticlestat 900 mg (Treatment C), Period 3: Placebo, (Treatment E), Period 4: Soticlestat 600 mg, (Treatment B), Period 5: Soticlestat 300 mg (Treatment A). Orally with a 7-day washout between doses.
- Treatment Phase, Sequence 7: EDACB: All participants received:
  Period 1: Placebo (Treatment E), Period 2: Alprazolam 2 mg (Treatment D), Period 3: Soticlestat 300 mg (Treatment A), Period 4: Soticlestat 900 mg (Treatment C), Period 5: Soticlestat 600 mg (Treatment B). Orally with a 7-day washout between doses.
- Treatment Phase, Sequence 8: AEBDC: All participants received:
  Period 1: Soticlestat 300 mg (Treatment A), Period 2: Placebo (Treatment E), Period 3: Soticlestat 600 mg (Treatment B), Period 4: Alprazolam 2 mg (Treatment D), Period 5: Soticlestat 900 mg (Treatment C). Orally with a 7-day washout between doses.
- Treatment Phase, Sequence 9: BACED: All participants received:
  Period 1: Soticlestat 600 mg (Treatment B), Period 2: Soticlestat 300 mg (Treatment A), Period 3: Soticlestat 900 mg (Treatment C), Period 4: Placebo (Treatment E), Period 5: Alprazolam 2 mg (Treatment D). Orally with a 7-day washout between doses.
- Treatment Phase, Sequence 10: CBDAE: All participants received:
  Period 1: Soticlestat 900 mg (Treatment C), Period 2: Soticlestat 600 mg (Treatment B), Period 3: Alprazolam 2 mg (Treatment D), Period 4: Soticlestat 300 mg (Treatment A), Period 5: Placebo (Treatment E). Orally with a 7-day washout between doses.
Period: Qualification Phase (3 Days)
Arm/Group | Qualification Phase: Sequence 1 | Qualification Phase: Sequence 2 | Treatment Phase, Sequence 1: ABECD | Treatment Phase, Sequence 2: BCADE | Treatment Phase, Sequence 3: CDBEA | Treatment Phase, Sequence 4: DECAB | Treatment Phase, Sequence 5: EADBC | Treatment Phase, Sequence 6: DCEBA | Treatment Phase, Sequence 7: EDACB | Treatment Phase, Sequence 8: AEBDC | Treatment Phase, Sequence 9: BACED | Treatment Phase, Sequence 10: CBDAE
Started | 50 | 50 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Qualification Safety Analysis Set (Treated) | 49 | 49 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 33 | 36 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 17 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did Not Meet Qualification Criteria | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Failure to Meet Continuation Criteria | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase (29 Days)
Arm/Group | Qualification Phase: Sequence 1 | Qualification Phase: Sequence 2 | Treatment Phase, Sequence 1: ABECD | Treatment Phase, Sequence 2: BCADE | Treatment Phase, Sequence 3: CDBEA | Treatment Phase, Sequence 4: DECAB | Treatment Phase, Sequence 5: EADBC | Treatment Phase, Sequence 6: DCEBA | Treatment Phase, Sequence 7: EDACB | Treatment Phase, Sequence 8: AEBDC | Treatment Phase, Sequence 9: BACED | Treatment Phase, Sequence 10: CBDAE
Started (Participants who completed Qualification Phase and met the qualification criteria were randomized to Treatment Phase. However, one participant was lost to follow-up after meeting the Qualification criteria and was not randomized in Treatment Phase.) | 0 | 0 | 7 | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 8 | 7
Safety Analysis Set (Treated) | 0 | 0 | 7 | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 7 | 7
Completed | 0 | 0 | 4 | 5 | 5 | 5 | 5 | 6 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 3 | 1 | 1 | 1 | 3 | 2 | 1 | 1 | 4 | 2
Not completed — Protocol Violation | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Qualification safety analysis set consists of all participants who received at least 1 dose of study drug in the qualification phase. As pre-specified in statistical analysis plan (SAP), the combined overall data for baseline measures were planned to be collected and reported for qualification phase.
Groups:
- Qualification Phase: All Participants: All participants who received at least 1 dose of study drug in the Qualification phase.:
  Sequence 1, Day 1: Alprazolam 2 mg, Day 2: Alprazolam matching placebo. Sequence 2, Day 1: Alprazolam matching placebo, Day 2: Alprazolam 2 mg. Orally with a 4-day washout between Qualification Phase and Treatment Phase.
Arm/Group | Qualification Phase: All Participants
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 90
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 74
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Phase: Drug Liking (Maximum Effect [Emax]) "At This Moment" as Assessed Using Bipolar Visual Analogue Scale (VAS)
Description: Drug liking ("at this moment") assessed how much a participant likes or dislikes a drug effect at the time the question was being asked. It was scored using a 0 to 100-point bipolar VAS, where 0: Strong disliking, 50: Neither like nor dislike (neutral point), 100: Strong liking. A higher score indicates stronger liking.
Time Frame: Day 1 of each Treatment Period: 15, 30, and 45 minutes, and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, and 24 hours post-dose
Population: The Modified Completer Analysis Set consisted of all participants in the Completer Analysis Set, excluding those whose Drug Liking "at this moment" VAS Emax scores met the elimination criteria defined in the SAP. As pre-specified in SAP, the pharmacodynamic data was planned to be collected and reported as per the treatment dose.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Treatment Phase: Soticlestat 300 mg: Soticlestat 300 mg as a single oral dose in one of five treatment periods.
- Treatment Phase: Soticlestat 600 mg: Soticlestat 600 mg as a single oral dose in one of five treatment periods.
- Treatment Phase: Soticlestat 900 mg: Soticlestat 900 mg as a single oral dose in one of five treatment periods.
- Treatment Phase: Alprazolam 2 mg: Alprazolam 2 mg as a single oral dose in one of five treatment periods.
- Treatment Phase: Placebo: Placebo as a single oral dose in one of five treatment periods.
Arm/Group | Treatment Phase: Soticlestat 300 mg | Treatment Phase: Soticlestat 600 mg | Treatment Phase: Soticlestat 900 mg | Treatment Phase: Alprazolam 2 mg | Treatment Phase: Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48
score on a scale | 56.7 (1.87) | 57.3 (1.89) | 56.5 (1.55) | 88.5 (1.58) | 55.6 (1.63)

2. Secondary Outcome: Treatment Phase: Overall Drug Liking (Emax) Assessed Using Bipolar VAS
Description: Overall drug liking assesses participant's overall experience with the drug by assessing the participant's overall liking for the drug. It was scored using a 100-point bipolar VAS, where 0: Strong disliking, 50: Neither like nor dislike (neutral point), 100: Strong liking. A higher score indicates better liking. The "overall drug liking" was an independent measure and not an "at this moment" assessment.
Time Frame: Day 1 of each Treatment Period: 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment Phase: Soticlestat 300 mg | Treatment Phase: Soticlestat 600 mg | Treatment Phase: Soticlestat 900 mg | Treatment Phase: Alprazolam 2 mg | Treatment Phase: Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48
score on a scale | 58.2 (2.40) | 58.5 (2.32) | 59.5 (2.45) | 90.0 (1.82) | 58.0 (2.17)

3. Secondary Outcome: Treatment Phase: Take Drug Again (Emax) Assessed "Overall" by Using Bipolar VAS
Description: Take drug again was a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It was scored using a 0 to 100-point bipolar VAS, where 0: Definitely not, 50: Neutral, 100: Definitely so. A higher score indicates stronger desire.
Time Frame: Day 1 of each Treatment Period: 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment Phase: Soticlestat 300 mg | Treatment Phase: Soticlestat 600 mg | Treatment Phase: Soticlestat 900 mg | Treatment Phase: Alprazolam 2 mg | Treatment Phase: Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48
score on a scale | 58.5 (2.80) | 57.6 (2.56) | 58.4 (2.72) | 92.0 (1.46) | 57.1 (2.14)

4. Secondary Outcome: Treatment Phase: Bad Drug Effects (Emax) Assessed "At This Moment" by Using Unipolar VAS
Description: Bad drug effects assessed the bad effect of drug experienced by the participant at the time the question is being asked. It was scored using a 100-point unipolar VAS, where responses were unidirectional and ranged from 0 (Not at all) to 100 (Extremely). A higher score indicated a stronger bad drug effect.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment Phase: Soticlestat 300 mg | Treatment Phase: Soticlestat 600 mg | Treatment Phase: Soticlestat 900 mg | Treatment Phase: Alprazolam 2 mg | Treatment Phase: Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48
score on a scale | 2.3 (1.58) | 1.4 (1.06) | 2.5 (2.08) | 28.5 (4.71) | 1.2 (0.93)

5. Secondary Outcome: Treatment Phase: Good Drug Effects (Emax) Assessed "At This Moment" by Using Unipolar VAS
Description: Good drug effects assessed the good effect of drug experienced by the participant at the time the question was being asked. It was scored using a 100-point unipolar VAS, where responses were unidirectional and range from 0 (Not at all) to 100 (extremely). A higher score indicated a stronger good drug effect.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment Phase: Soticlestat 300 mg | Treatment Phase: Soticlestat 600 mg | Treatment Phase: Soticlestat 900 mg | Treatment Phase: Alprazolam 2 mg | Treatment Phase: Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48
score on a scale | 10.9 (3.18) | 10.1 (2.78) | 11.6 (3.10) | 74.0 (3.42) | 8.1 (2.74)

6. Secondary Outcome: Treatment Phase: High (Emax) Assessed "At This Moment" by Using Unipolar VAS
Description: High assessed the degree that a participant feels a good effect (that is, euphoria) at the time the question was being asked. It was scored using a 100-point unipolar VAS, where responses were unidirectional and ranged from 0 (Not at all) to 100 (Extremely). A higher score indicated a stronger high effect.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment Phase: Soticlestat 300 mg | Treatment Phase: Soticlestat 600 mg | Treatment Phase: Soticlestat 900 mg | Treatment Phase: Alprazolam 2 mg | Treatment Phase: Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48
score on a scale | 10.3 (2.95) | 12.0 (2.94) | 11.3 (3.16) | 72.8 (3.49) | 8.1 (2.62)

7. Secondary Outcome: Treatment Phase: Number of Participants With One or More Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE was defined as an adverse event that started or worsened during or after the first dose of study drug.
Time Frame: From start of study drug administration (Day 1) up to Day 37
Population: The Safety Analysis Set consisted of all participants who received at least 1 dose of study drug in the Treatment phase. As pre-specified in SAP, the safety data was planned to be collected and reported as per treatment dose. Here, "overall number of participants analyzed" signified participants who received the specified treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Phase: Soticlestat 300 mg | Treatment Phase: Soticlestat 600 mg | Treatment Phase: Soticlestat 900 mg | Treatment Phase: Alprazolam 2 mg | Treatment Phase: Placebo
Number analyzed (Participants) | 63 | 63 | 61 | 59 | 62
Participants | 17 | 12 | 13 | 52 | 15

ADVERSE EVENTS:
Time Frame: TEAEs are AEs that started after the first dose of study drug administration (Day 1) up to Day 3 for Qualification Phase and up to Day 37 for Treatment Phase
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. As pre-specified in SAP, the safety data was planned to be collected and reported as per treatment dose. Here, participants "at Risk" signified participants who received the specified treatment.
Groups:
- Qualification Phase: Placebo: Alprazolam matching placebo orally, once on Day 1 or once on Day 2 in Qualification Phase.
- Qualification Phase: Alprazolam 2 mg: Alprazolam 2 mg, orally, once on Day 1 or once on Day 2 in Qualification Phase.
Arm/Group | Qualification Phase: Placebo | Qualification Phase: Alprazolam 2 mg | Treatment Phase: Soticlestat 300 mg | Treatment Phase: Soticlestat 600 mg | Treatment Phase: Soticlestat 900 mg | Treatment Phase: Alprazolam 2 mg | Treatment Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/98 | 0/63 | 0/63 | 0/61 | 0/59 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/98 | 0/63 | 0/63 | 0/61 | 0/59 | 0/62
Other Adverse Events (participants affected / at risk) | 2/96 | 83/98 | 14/63 | 10/63 | 9/61 | 50/59 | 8/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Qualification Phase: Placebo (N=96) | Qualification Phase: Alprazolam 2 mg (N=98) | Treatment Phase: Soticlestat 300 mg (N=63) | Treatment Phase: Soticlestat 600 mg (N=63) | Treatment Phase: Soticlestat 900 mg (N=61) | Treatment Phase: Alprazolam 2 mg (N=59) | Treatment Phase: Placebo (N=62)
Headache (Nervous system disorders) | 0 | 1 | 4 | 1 | 2 | 4 | 1
Somnolence (Nervous system disorders) | 2 | 73 | 9 | 6 | 3 | 44 | 6
Euphoric mood (Psychiatric disorders) | 0 | 26 | 1 | 5 | 4 | 23 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT05602818/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT05602818/SAP_001.pdf